CLINICAL TRIAL: NCT01896063
Title: EA Induces Sedative and Hypnotic Effects by Detecting BIS Value and MRI.
Brief Title: Sedative and Hypnotic Effects Induced by EA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, wangqiang, Department of anesthesijology, Xijing Hospital
Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: wangqiang888
Record Dates: First submitted 2013-01-07; First posted 2013-07-11 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Bypass Complications
Keywords: Electroacupuncture, Sedation
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Electroacupuncture preconditioning (Experimental)
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture

SUMMARY:
Insomnia is a common clinical disease.The serious patients could not sleep all night, often accompanied by headache, dizziness, forgetfulness and so on. All of these increase the mental burden of insomnia patients and seriously affected the normal work and quality of life of patients. Modern medical treatment to treat insomnia is using sedative and hypnotic drugs, mainly benzodiazepine, zopiclone. But long-term use of these drugs can induce the adverse reactions, including resistance, dependence and addiction. Many articles indicate that electroacupuncture can effectively improve insomnia, play the role of sedative and hypnotic effect and avoid many adverse reactions and side effects. Then there are no more objective indicators to affirm that which part of brain takes place the appropriate changes when electroacupuncture induces the sedative effect. So we designed this experiment.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to go with EA
* Can not have any disease

Exclusion Criteria:

* Overworked recently

Ages: 24 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
BIS value | 30 minutes
  The primary outcome is assessing whether BIS value reduce during electroacupuncture stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Wang, Dr., Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Lu Z, Huo T, Deng J, Guo F, Liu K, Liu P, Wang Q, Xiong L. Transcutaneous electrical acupoint stimulation induced sedative effects in healthy volunteers: A resting-state fMRI study. Front Hum Neurosci. 2023 Jan 19;16:843186. doi: 10.3389/fnhum.2022.843186. eCollection 2022. PMID 36741778